CLINICAL TRIAL: NCT06858540
Title: A Blended Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Chinese Adolescents With Non-suicidal Self-injury: A Pilot Study
Brief Title: Blended Unified Protocol in Chinese Adolescents With Non-Suicidal Self-Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Jun Ou (Other)
Responsible Party: Sponsor-Investigator, Jian-Jun Ou, Principal Investigator, Central South University
Organization: Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2024203
Record Dates: First submitted 2025-02-26; First posted 2025-03-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-02

CONDITIONS: Non-suicidal Self-injury (NSSI)
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants will receive an 8-week blended version of the Unified Protocol for Adolescents.
  Interventions: Behavioral: Unified protocol for transdiagnostic treatment of emotional disorders in adolescents

INTERVENTIONS:
Behavioral: Unified protocol for transdiagnostic treatment of emotional disorders in adolescents — The blended UP-A includes 8 weekly modules, 6 of which (Module 2 - 7)are online self-guided sessions. The online self-guided sessions will last approximately 45 minutes each. Over the course of these 6 weeks, participants will also have 6 therapist-guided online sessions via videoconference, each lasting 30 minutes. Two face-to-face individual sessions are scheduled, one at the beginning of each (Module 1) and one at the end (module 8), each with an expected duration of 90 minutes.

SUMMARY:
This study utilizes the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) to address non-suicidal self-injury among Chinese adolescents. This program is an annualized cognitive-behavioral therapy designed for adolescents aged 12-17 years who engage in non-suicidal self-injury behavior. Its primary goal is to reduce the intensity and frequency of distressing emotional experiences by teaching adolescents how to confront and respond to these emotions in more adaptive ways. In turn, this helps reduce self-injury impulses and behaviors. The UP-A is adapted to the Chinese cultural context and delivered as a blended treatment, combining face-to-face and online sessions. The study will assess the feasibility, acceptability, and preliminary efficacy of this intervention through a single-arm design, which includes pretest, posttest, and follow-up assessments.

DETAILED DESCRIPTION:
The blended UP-A includes 8 weekly modules, 6 of which (Module 2 - 7)are online self-guided sessions. The online self-guided sessions will last approximately 45 minutes each. Over the course of these 6 weeks, participants will also have 6 therapist-guided online sessions via videoconference, each lasting 30 minutes. Two face-to-face individual sessions are scheduled, one at the beginning of each (Module 1) and one at the end (module 8), each with an expected duration of 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 12 and 17 years;
2. Engaged in non-suicidal self-injury (NSSI) at least 5 times in the past 12 months, with at least 1 episode in the past month;
3. Minimum education level of primary school or above;
4. Participant and guardian fully understand the research content and agree to participate, with signed informed consent provided.

Exclusion Criteria:

1. Suicide attempts in the past month or a score of ≥17 on the MINI National Neuropsychiatric Interview for Children (MINI KID 5.0), indicating a high risk of suicide;
2. Diagnosis of a psychotic disorder, manic or hypomanic episode, autism spectrum disorder, or other serious neurodevelopmental disorders according to the DSM-5;
3. Presence of severe physical illness or other medical conditions that may affect the completion of treatment and evaluation;
4. Currently receiving other professional psychotherapy or participating in another NSSI intervention study;
5. Received 5 or more sessions of cognitive behavioral therapy (CBT) in the past 5 years;
6. Having received electroconvulsive therapy (ECT) within the past 6 months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | Immediately after the intervention
  Adherence to the intervention will be measured by the number of sessions attended and the number of participants who complete at least 70% of the sessions, the timing of these sessions (within the designated week or not), the number of interactive exercises completed in each session, and the completion of home assignment tasks.
Dropout rates | Immediately after the intervention
  Dropout rates are defined as the number of participants who dropped out from the intervention before completing it.
The Feasibility and Acceptability Questionnaire (FAQ) | Immediately after the intervention
  The FAQ will be used to evaluate the feasibility and acceptability of the intervention. The FAQ consists of three subscales, each containing six items: (1) experience using the online platform, (2) satisfaction with the program, (3) therapeutic alliance. The higher scores indicate greater feasibility and acceptability.
Participants' perspectives on the intervention | Immediately after the intervention
  Participants' perspectives on the intervention will be assessed through semi-structured interviews, exploring the factors that facilitate or hinder their adherence to and completion of the program.

SECONDARY OUTCOMES:
Non-suicidal self-injury | baseline, immediately after the intervention, and 1-month after the intervention
  The Adolescent Self-Harm Behavior Scale includes 18 items describing forms of self-harm. The scale is divided into two dimensions: frequency and severity of self-harm. Self-harm frequency is scored on a 4-point scale (0-3), with the following categories: 0 times, 1 time, 2-4 times, and more than 5 times. The severity of physical injury is scored on a 5-point scale (0-4), with the following categories: none, mild, moderate, severe, and extremely severe. The product of frequency and injury severity for each item is used as the overall score for NSSI, with higher scores indicating more severe NSSI behavior.
Emotion dysregulation | baseline, immediately after the intervention, and 1-month after the intervention
  Difficulties in Emotion Regulation Scale (DERS) is used to assess the participants' emotional regulation abilities. It consists of 36 items across 6 dimensions, with higher total scores indicating a higher level of emotional dysregulation. The dimensions include: emotional awareness, emotional acceptance, impulse control, emotional understanding, goal-directed behavior, and strategy use.
Emotion regulation strategies | baseline, immediately after the intervention, and 1-month after the intervention
  The Emotion Regulation Questionnaire (ERQ) is used to measure participants' emotional regulation strategies. It consists of 10 items, divided into two dimensions: cognitive reappraisal and expressive suppression. Each item is rated on a 7-point scale, with higher scores indicating a stronger tendency to use the corresponding emotional regulation strategy.
Depression | baseline, immediately after the intervention, and 1-month after the intervention
  The Patient Health Questionnaire-9 (PHQ-9) was used to measure depression levels. This nine-item scale rates each item on a four-point scale from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 27. Higher scores indicate greater depression severity.
Anxiety | baseline, immediately after the intervention, and 1-month after the intervention
  The Generalized Anxiety Disorder-7 (GAD-7) was used to assess anxiety levels of participants. This seven-item scale also employs a four-point scoring system from 0 ("not at all") to 3 ("nearly every day"), with higher scores reflecting greater anxiety severity.

OTHER OUTCOMES:
Basic psychological need satisfaction and frustration | baseline, immediately after the intervention, and 1-month after the intervention
  The Basic Psychological Need Satisfaction and Frustration Scale (BPNSF) was developed by Chen in 2015. The scale consists of two subscales: basic psychological need satisfaction and basic psychological frustration. The Basic Psychological Need Satisfaction subscale includes three dimensions-autonomy satisfaction, competence satisfaction, and relatedness satisfaction-comprising 12 items in total. The Basic Psychological Need Frustration subscale includes three dimensions-autonomy frustration, competence frustration, and relatedness frustration-also comprising 12 items. Participants are asked to rate each item on a 5-point Likert scale (1 = Strongly Disagree; 5 = Strongly Agree).
Neuroticism | baseline, immediately after the intervention, and 1-month after the intervention
  The Neuroticism subscale from the Neuroticism-Extraversion-Openness Five-Factor Inventory was selected to measure neuroticism. The Neuroticism subscale consists of 12 items, rated on a 5-point Likert scale. Higher scores indicate a stronger tendency toward neuroticism in the individual.
Distress tolerance | baseline, immediately after the intervention, and 1-month after the intervention
  The Distress Tolerance Scale (DTS) is a 15-item measure of an individual's perceived ability to withstand negative emotions. Items are answered on a five-point Likert scale ranging from 1 = strongly agree to 5 = strongly disagree. Traditionally, high DTS-global distress intolerance scores reflect a heightened ability to tolerate distress, whereas low total scores represent distress intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No